CLINICAL TRIAL: NCT04853875
Title: Visiting Staff, Division of Gastroenterology and Department of Internal Medicine, Mackay Memorial Hospital, Taipei, Taiwan
Brief Title: ILTHPI - Comparison of Medicament Containing Tetracycline, Metronidazole, Bismuth Versus Amoxicillin, Metronidazole, Clarithromycin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Principal Investigator, Tai-cherng Liou, MD, Principle investigator, Mackay Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21MMHIS016e
Record Dates: First submitted 2021-04-14; First posted 2021-04-21 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter Pylori; Proton pump inhibitor; Amoxicillin; Metronidazole; Bismuth; Tetracycline; Clarithromycin
MeSH Terms: interventions — Tetracycline; Metronidazole; bismuth tripotassium dicitrate; bismuth oxide; Amoxicillin; Clarithromycin

STUDY DESIGN:
Intervention Model Description: 104 participants are randomly assigned to receive intraluminal eradication of H. pylori.
  with medicaments containing Tetracycline, Metronidazole, and Bismuth versus Amoxicillin, Metronidazole, and Clarithromycin.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Tetracycline, Metronidazole, and Bismuth) (Experimental): Intraluminal Therapy for Helicobacter pylori Infection - Single dose medicament containing Tetracycline 2g, Metronidazole 2g, and Bismuth subcitrate 480 mg
  Interventions: Drug: Tetracycline, Metronidazole, Bismuth subcitrate
- Group B (Amoxicillin, Metronidazole, and Clarithromycin) (Active Comparator): Intraluminal Therapy for Helicobacter pylori Infection - Single dose medicament containing Amoxicillin 3g, Metronidazole 2g, and Clarithromycin 1g
  Interventions: Drug: Amoxicillin, Metronidazole, Clarithromycin

INTERVENTIONS:
Drug: Tetracycline, Metronidazole, Bismuth subcitrate — 52 participants (Group A) are randomly assigned to receive intraluminal eradication of H. pylori with medicament containing Tetracycline, Metronidazole, and Bismuth subcitrate
  Other Names: Bismuth Trioxide
  Arms: Group A (Tetracycline, Metronidazole, and Bismuth)
Drug: Amoxicillin, Metronidazole, Clarithromycin — 52 participants (Group B) are randomly assigned to receive intraluminal eradication of H. pylori with medicament containing Amoxicillin, Metronidazole, and Clarithromycin
  Other Names: Klaricid
  Arms: Group B (Amoxicillin, Metronidazole, and Clarithromycin)

SUMMARY:
Helicobacter pylori (H. pylori) is a spiral shaped, microaerophilic, gram negative bacterium. The organism resides in the acid and mucous layer of the human gastric mucosa, adheres to and colonizes the mucosal surface of the stomach and the mucosal epithelium with gastric metaplasia of duodenal bulb. Many studies have shown that H. pylori is an important causal factor of chronic gastritis, peptic ulcer disease, gastric cancer and gastric lymphoma. Endoscopic examination is indicated to confirm the above diagnosis for patient with H. pylori infection. The eradication rate of standard triple therapy has fallen below 80% in many countries due to the worldwide increasing prevalence of antibiotic resistant strains. This is related to the special gastric milieu of H. pylori, which leads to a more difficult and complicated treatment for achieving a successful eradication rate than other bacteria. Several strategies have been proposed to increase the eradication rate in the first line therapy or as a rescue therapy. However, these rescue therapies will increase the side effects and costs of treatment, decrease the compliance of patients and increase the rate of worldwide antibiotic resistance steadily. The WHO has listed H. Pylori as one of 12 antibiotic-resistant bacteria that have the greatest threat to human health in Feb. 2017. Our previous studies suggested that the administration of single -dose therapeutic agents can achieve the eradication of H. pylori immediately while conducting the endoscopic examination. The eradication rate of intraluminal therapy for H. pylori infection (ILTHPI) is 53.7% (51/95), and control the intragastric pH above 4 prior to the ILTHPI can even reach a 72.0%(36/50) eradication rate of H. pylori.

According to the recent Taiwan consensus for the treatment of H. pylori in 2017, the first line therapeutic regiment of H. pylori containing Amoxicillin, Clarithromycin, and Metronidazole if the rate of Clarithromycin resistance is below 15%, while the first line therapeutic regiment of H. pylori containing tetracycline, metronidazole, and bismuth subcitrate if the rate of Clarithromycin resistance is above 15%. We aimed to evaluate and compare the efficacy of medicament containing Tetracycline, Metronidazole, and Bismuth versus Amoxicillin, Metronidazole, and Clarithromycin for the Intraluminal therapy of Helicobacter pylori infection.

DETAILED DESCRIPTION:
During the endoscopic examination, patient is sedated with intravenous Midazolam 5mg and Fentanyl 0.05mg, the vital signs will be closely monitored by physiological monitor (PHILIPS SureSigns VM6). The treatment will be terminated immediately if unstable vital sign detected or if patient asks for termination. The pH value of gastric juice will be measured with the pH test strips. and the he gastric mucus is irrigated with acetylcysteine solution. The investigators randomly assigned medicaments containing different antibiotic powders either Tetracycline 2g, Metronidazole 2g, and Bismuth 480mg (Group A) or Amoxicillin 3g, Metronidazole 2g, and Clarithromycin 1g (Group B) to dispense on the surface of gastric mucosa and duodenal mucosa of duodenal bulb. After the intraluminal therapy, patients will rest for 30 to 60 minutes and go home if the effect of sedation subsided. Patients can take meal if no abdominal discomfort. C13-Urea breath test (UBT) will be used to assess the existence of H. pylori 2 weeks after the intraluminal therapy. Patients failed to achieve intraluminal eradication of H. pylori will be assigned to 7-day concomitant therapy (Group A) or 7-day bismuth quadruple therapy (Group B). The C13-UBT will be used to assess the existence of H. pylori 4 weeks after the oral antibiotic therapy. The overall eradication rates of the intraluminal therapy plus the oral antibiotics therapies will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged between 20 years and 75 years
2. Patients have H. pylori infection and have not treated with oral antibiotics
3. Patients are willing to receive the intraluminal therapy. The written informed consents will be obtained from all patients prior to enrollment.

Exclusion Criteria:

* Patients will be excluded from the study if any one of the following criteria is present:

  1. Children and teenagers aged less than 20 years, or adult greater than 75 years
  2. Contraindication for endoscopic examination or food retention in the gastric lumen
  3. History of gastrectomy; Gastroduodenal stenosis、deformity or obstruction; Gastroduodenal malignancy, including adenocarcinoma and lymphoma
  4. Contraindication to treatment drugs: previous allergic reaction to antibiotics of study, PPI (Lansoprazole), Acetylcysteine and Sucralfate; pregnant or lactating women
  5. Severe concurrent acute or chronic illness: renal failure, decompensated cirrhosis of liver, incurable malignant disease
  6. Patients who cannot give informed consent by himself or herself

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-12-16 (Actual)

PRIMARY OUTCOMES:
The eradication rates of intraluminal therapy | C13-UBT will be used to assess the existence of H. pylori 2 weeks after the intraluminal therapy
  To evaluate and compare the eradication rates of different medicaments for the Intraluminal Therapy for Helicobacter pylori Infection between Group A and Group B.

SECONDARY OUTCOMES:
The adverse events of intraluminal therapy | Within one week after the Intraluminal Therapy for Helicobacter pylori Infection
  of different medicaments for the Intraluminal Therapy for Helicobacter pylori Infection between Group A and Group B.
The eradication rates of oral antibiotic rescue therapies | C13-UBT will be used to assess the existence of H. pylori 4 weeks after the oral antibiotics rescue therapy
  To evaluate and compare the eradication rates of different oral antibiotic rescue therapies for failed Intraluminal Therapy between concomitant therapy ( Group A) and bismuth-based quadruple therapy (Group B)
The adverse events of oral antibiotic rescue therapies | Within one week after complete the oral antibiotics rescue therapy
  To evaluate and compare the adverse events of different oral antibiotic rescue therapies for failed Intraluminal Therapy between concomitant therapy ( Group A) and bismuth-based quadruple therapy (Group B)

CONTACTS AND LOCATIONS:
Overall Officials: Tai-cherng Liou, MD, Principal Investigator — Division of Gastroenterology and Department of Internal Medicine, Mackay Memorial Hospital
Locations (1):
- Division of Gastroenterology and Department of Internal Medicine, Mackay Memorial Hospital, Taipei, Taiwan